CLINICAL TRIAL: NCT05144308
Title: Assessment of Visual and Refractive Results, and Rotational Stability of the TECNIS® Eyhance Toric II 1-piece Posterior Chamber Lens in Patients With Astigmatism Undergoing Cataract Surgery: a Prospective Cohort Study - STATE
Brief Title: Assessment of Visual and Refractive Results and Rotational Stability of the TECNIS® Eyhance Toric II 1-piece Posterior Chamber Lens in Patients With Astigmatism Undergoing Cataract Surgery
Acronym: STATE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor-investigator agreement
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JFO_2021_10
Record Dates: First submitted 2021-11-10; First posted 2021-12-03 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Cataract; Astigmatism
Keywords: TECNIS® Eyhance Toric II 1-piece posterior chamber lens
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Intervention Model Description: Single-center prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients operated with a TECNIS® Eyhance Toric II 1-piece posterior chamber lens (Experimental): For at least one eye : Planned cataract surgery with placement of a TECNIS® Eyhance Toric II 1-piece posterior chamber lens
  Interventions: Procedure: Images of the operated eye (s)

INTERVENTIONS:
Procedure: Images of the operated eye (s) — Through the operating microscope or a slit lamp, dilated pupil. Taken on the day of surgery (D0) and at 1 week, 1 month and 3 months post-op

SUMMARY:
Cataract surgery is one of the most common procedures performed worldwide. Astigmatism is the most common refractive disorder in adults, hence there is a high prevalence of preexisting astigmatism in cataract patients. Access to astigmatism correction during cataract surgery allows for improved visual outcomes for patients. Toric intraocular lenses (IOLs) are the procedure of choice to correct corneal astigmatism of one diopter or more in cases undergoing cataract surgery. Rotational stability is a key factor for successful outcomes with toric IOLs. Postoperative toric IOL misalignment is the major factor responsible for suboptimal visual outcomes after toric IOL implantation.

The TECNIS® Eyhance Toric II 1-piece posterior chamber lens is a new toric IOL which is FDA approved and CE marked. Marketed by Johnson & Johnson Vision, it is indicated for the visual correction of aphakia and pre-existing corneal astigmatism of one diopter or greater in adult patients with or without presbyopia in whom a cataractous lens has been removed by phacoemulsification and who desire reduction in residual refractive cylinder.

No study assessing the early rotational stability of the TECNIS® Eyhance Toric II IOL has been published yet.

ELIGIBILITY:
Inclusion criteria

* Aged ≥ 18 years
* Patients scheduled for bilateral cataract surgery
* For at least one eye :

  * Cataract surgery clinically indicated
  * Corneal astigmatism ≥ 1 D
  * Planned cataract surgery with placement of a TECNIS® Eyhance Toric II 1-piece posterior chamber lens

Non inclusion criteria

* Pregnant or breast-feeding women
* In the eye with planned cataract surgery with placement of a TECNIS® Eyhance Toric II 1-piece posterior chamber lens:

  * Irregular astigmatism (keratoconus suspicion)
  * Corneal scaring in visual axis
  * Retinal impairment that may limit visual recovery (macular degeneration, history of retinal detachment, etc.)
  * Visually impaired eye since childhood that cannot be improved despite correction of the refractive disorder
  * Any other ophthalmic disease inducing visual impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-10-09 (Actual)

PRIMARY OUTCOMES:
The mean of the best monocular uncorrected distance visual acuity UDVA (logMAR) at 1 month post-operative | 1 month
The mean of the best monocular corrected distance visual acuity (CDVA) (logMAR) preoperative (maximum 12 months before surgery) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc FEBBRARO, MD, Principal Investigator — Hôpital Fondation A. de Rothschild
Locations (1):
- Hôpital Fondation A. de Rothschuld, Paris, Hôpital Fondation A. de Rothschild, France